CLINICAL TRIAL: NCT05812885
Title: Transcutaneous Electrical Nerve Stimulation (TENS) and Chronic Low-Back Pain: A Randomized Crossover Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) and Low Back Pain
Acronym: TENS and LBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Principal Investigator, Richard Liebano, Associate Professor, University of Hartford
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23-03-187
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active TENS (Experimental): Active TENS: 100 Hz, 200 μs at maximal tolerable intensity
  Interventions: Device: TENS
- Placebo TENS (Placebo Comparator): Placebo TENS: 100 Hz, 200 μs on for 45 seconds and then ramps off.
  Interventions: Device: TENS
- No TENS (No Intervention): Participants will wear a TENS unit that will be turned off to blind the outcome assessor

INTERVENTIONS:
Device: TENS — Active TENS
  Arms: Active TENS; Placebo TENS

SUMMARY:
Low back pain is a significant public health problem, is very prevalent, and is often characterized by the persistence of symptoms. Unfortunately, substantial improvements in people with chronic low back pain are rare, causing most people to live with the pain. People with chronic low back pain may have an exaggerated pain response to nociceptive input into tissues that may also cause symptoms distant from the site of the primary symptoms. Historically, these symptoms were thought to be related to pathoanatomic changes to the muscles, ligaments, or joints. However, the severity of these structural changes weakly correlates with the clinical presentation and, in most cases, is not directly related to diagnostic image findings. Patients with chronic musculoskeletal pain, in general, show signs of local/central sensitization. The central sensitization may appear to be directly correlated with the intensity and duration of pain. Therefore, it is essential to reduce pain intensity and minimize the duration of pain to prevent this from happening.

Pain relief for chronic low back pain patients should be aimed at treatments that reduce central excitability and increase central inhibition. Research into chronic low back pain treatment has demonstrated strong evidence that different types of exercise decrease pain and improve quality of life. However, exercise itself may be painful, preventing a person from exercising. Thus, treatments aimed at decreasing pain will improve a person's ability to exercise and participate in activities of daily living.

One treatment aimed at reducing central excitability and increasing central inhibition is transcutaneous electrical nerve stimulation (TENS). TENS is a "non-pharmacological" treatment for pain that is inexpensive, safe, and easy to use. Prior studies show that TENS utilizes opioid receptors both spinally and supraspinally to inhibit nociceptive dorsal horn neurons, reduce excitatory neurotransmitter release, and reduce hyperalgesia. Thus, TENS may be particularly useful in people with chronic low back pain because it can activate descending inhibitory pathways (reduced in chronic low back pain patients) and inhibit central excitability (increased in chronic low back pain patients).

Previous studies that have investigated the effects of TENS on pain in low back pain patients have failed to use proper intensities of current, and the assessment of pain was not performed during the peak of the analgesic response. Previous studies show inadequate intensities do not reduce pain or increase pressure pain thresholds. Further, TENS typically does not affect resting pain, while changes in pressure pain thresholds and pain with movement are reduced. Thus, the current study proposes to assess the effects of TENS on measures of pain, function, and descending inhibition using the maximal tolerable intensity of TENS applied to a large area of the trunk.

DETAILED DESCRIPTION:
The study will be a simple crossover design with the following three treatments (1) active TENS, (2) placebo TENS or (3) no treatment control randomly assigned. Each subject will receive all 3 interventions in random order.

The following tools will be used to measure pain (Numeric Rating Scale), central excitability (pressure pain thresholds, temporal summation and CPM) and function (sit-to-stand test and repeated trunk flexion).

ELIGIBILITY:
Inclusion Criteria:

* people who have experienced back pain for at least 3 months
* and have reported a minimal pain level of 3 on the 0-10 Pain Numerical Rating Scale (NRS)
* age from 18-60
* TENS naive or have not used TENS for 5 years.
* Both men and women may participate in the study

Exclusion Criteria:

* Serious spinal disorders, such as fractures, tumors, or inflammatory arthritis disease
* nerve root disorders confirmed by neurological tests;
* neurological diseases
* severe cardiorespiratory disease
* pregnancy
* skin infection or lesions or change in sensation at the TENS application site
* cancer
* cardiac pacemaker
* allergy to electrodes
* use of opioids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Pain at Rest | 3 weeks
  Pain at Rest Difference Score Pre-intervention and Post Intervention measured by the Numeric Pain Rating Scale. It starts with the absence of pain (0) and reaches the worst pain imaginable (10).
Pain With Movement | 3 weeks
  Pain With Movement Difference Score Pre-intervention and Post Intervention measured by the Numeric Pain Rating Scale. It starts with the absence of pain (0) and reaches the worst pain imaginable (10).

SECONDARY OUTCOMES:
Sit-to-Stand Test | 3 weeks
  Five sit-to-stand repetitions will be completed in two trials with an average of two trials for scoring
Repeated trunk flexion | 3 weeks
  From a neutral standing position, the subject will be required to flex to the limit of the range and return to the upright position as fast as tolerable.This activity will be repeated 10 times, and the total procedure will be timed with a stopwatch
Pressure Pain Threshold (PPT) | 3 weeks
  A digital pressure algometer will measure the pain threshold to deep mechanical stimuli.
Heat Pain Threshold (HPT) | 3 weeks
  Superficial heat pain sensitivity will be assessed using a handheld thermode.
Temporal Summation | 3 weeks
  Temporal summation will be induced by a pressure algometer
Conditioned pain modulation | 3 weeks
  A cold pressor test will be used to assess the activation of the conditioned pain modulation.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, PhD, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liebano RE, Sluka KA, Roy J, Savinelli M, Dailey DL, Riley SP. Effects of transcutaneous electrical nerve stimulation on pain, function, and descending inhibition in people with non-specific chronic low-back pain: a study protocol for a randomized crossover trial. Trials. 2024 Apr 6;25(1):242. doi: 10.1186/s13063-024-08089-7. PMID 38582874